CLINICAL TRIAL: NCT06671600
Title: Effects of Osteopathic Manipulative Treatment Protocol on Sleep Quality in Parkinson's Disease Subjects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYIT IRB-2025-158
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Parkinsons Disease; Sleep
Keywords: OMM; Sleep; Parkinsons Disease; Osteopathy
MeSH Terms: conditions — Parkinson Disease | interventions — Manipulation, Osteopathic; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into either the treatment group who will receive OMT and the sham group who will receive light touch.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (OMT) (Experimental): For the Osteopathic Manipulative Medicine(OMM) treatment group, an osteopathic manipulative treatment protocol will be applied to the cranial, cervical, thoracic, and ribcage regions. OMM procedures performed on the treatment group will consist of
  1. suboccipital decompression/release
  2. base spread
  3. occipitoatlantal (OA) decompression
  4. venous sinus drainage
  5. compression of the fourth ventricle
  6. cervical myofascial (unilateralperpendicular stretch)
  7. thoracic inlet release (direct or indirect)
  8. Bilateral rib raising
  9. thoracoabdominal diaphragm doming (direct technique)
  10. pedal pump (Dalrymple lymphatic pump). All aforementioned techniques are based on the protocol from Foundations of Osteopathic Medicine.
  Interventions: Procedure: Osteopathic Manipulative Treatment
- Sham- light touch (Sham Comparator): The sham group will serve as the control group and will receive a light touch-control procedure based on prior study utilizing light touch
  Interventions: Procedure: Sham (No Treatment)

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — Osteopathic manipulative treatment(OMT) protocol will be applied to the cranial, cervical, thoracic, and ribcage regions. OMT procedures performed on the treatment group will consist of
  1. suboccipital decompression/release
  2. base spread
  3. occipitoatlantal (OA) decompression
  4. venous sinus drainage
  5. compression of the fourth ventricle
  6. cervical myofascial (unilateral perpendicular stretch)
  7. thoracic inlet release (direct or indirect)
  8. Bilateral rib raising
  9. thoracoabdominal diaphragm doming (direct technique)
  10. pedal pump (Dalrymple lymphatic pump)
  Arms: Treatment Group (OMT)
Procedure: Sham (No Treatment) — The sham group will serve as the control group and will receive a light touch-control procedure based on prior study utilizing light touch.
  Arms: Sham- light touch

SUMMARY:
Parkinsonism, mainly caused by Parkinsons disease (PD), includes symptoms like tremors, stiffness, slow movements, and balance problems. These symptoms can make it hard for people to sleep well, which leads to a lower quality of life and can increase the risk of other health issues and cognitive decline.

Osteopathic manipulative treatment (OMT) is a hands-on approach that may help improve sleep without the side effects of traditional treatments. While OMT has shown promise in enhancing sleep, no studies have specifically looked at its effects on sleep in Parkinson's disease patients.

This study aims to see if OMT can help improve sleep quality, cognitive function, and daily activities for people with PD. The investigators will focus on treating specific areas of the body, using techniques that have helped improve sleep in the past.

Participants will be divided into two groups: one will receive OMT, while the other will get a light touch treatment as a control. Sleep surveys and data from Fitbit devices will be used to compare the effects of the two treatments. Additionally, cognitive function will be assessed using a specific task called the Stroop task.

This research could show that OMT can be a valuable addition to treatments for improving sleep quality in people with Parkinsons disease.

DETAILED DESCRIPTION:
Parkinsonism is primarily linked to Parkinsons disease (PD) and presents a range of symptoms including tremors at rest, muscle stiffness, slowed movement (bradykinesia), and difficulties with balance. These symptoms can significantly disrupt sleep patterns, making it challenging for individuals to both fall asleep and stay asleep. As a result, many patients experience reduced sleep quality, which can adversely affect their overall well-being and make them more vulnerable to additional health problems, including cognitive decline.

Osteopathic manipulative treatment (OMT) is a holistic, hands-on therapy aimed at enhancing the body's natural ability to heal and function. It focuses on manipulating the body's muscles and joints to improve circulation and promote relaxation, which may lead to better sleep outcomes. Unlike some conventional treatments that often come with unwanted side effects, OMT offers a potentially safer, individualized approach to managing sleep disorders, especially in the context of Parkinsons disease.

Despite the promising indications that OMT could improve sleep quality, there has been a lack of focused research on its application specifically for patients with Parkinsons disease. This study aims to fill that gap by investigating how targeted OMT can influence sleep quality, cognitive function, and daily activities in individuals diagnosed with PD.

The treatment protocol will specifically target areas of the body such as the cranial, cervical, thoracic, and rib regions, using established OMT techniques that have previously shown efficacy in enhancing sleep quality. Participants will be assigned to one of two groups: the treatment group receiving OMT and a control group receiving a light touch treatment, which serves as a placebo.

To assess the effectiveness of the OMT, the investigators will employ a variety of measurement tools. Sleep quality will be evaluated through self-reported surveys as well as objective data collected using Fitbit devices, which can track sleep patterns and quality metrics. Additionally, cognitive function, particularly executive function, will be assessed through the Stroop task, a well-established cognitive test that measures a persons ability to manage conflicting information.

By systematically comparing the outcomes of the OMT group to those of the control group, this research aims to demonstrate the potential benefits of OMT as a complementary treatment for improving sleep quality in patients with Parkinsons disease. The findings could pave the way for integrating OMT into standard care practices, ultimately enhancing the quality of life for individuals living with this challenging condition.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of Parkinson's disease as per a neurologist
* Severity of 0-3 on the Hoehn and Yahr (H-Y) Scale
* Able to receive OMM
* Able to be in a supine and prone position.
* Able to wear a Fitbit watch and an oxygen saturation ring for the duration of the study (including when sleeping).
* Have sleep disturbance complaints.

Exclusion Criteria:

* Patients on medications that affect sleep
* Have a pre-existing sleep disorder diagnosis
* Those who have a concurrent neurological diagnosis that would confound sleep patterns (ie. narcolepsy)
* Contraindications to the OMM techniques used in this protocol
* Severity of 4 and 5 on the Hoehn and Yahr Scale

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-08 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | 5 weeks
  Heart rate will be measured with a Fitbit watch
Sleep quality | 5 weeks
  sleep quality will be measured using a Fitbit device
Sleep duration | 5 weeks
  Sleep duration will be measured using a Fitbit device
Oxygen saturation | 5 weeks
  Oxygen saturation will be measured using a Fitbit device
Sleep stage | 5 weeks
  Time in each sleep stage will be recorded using FitBit

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hablitz LM, Nedergaard M. The Glymphatic System: A Novel Component of Fundamental Neurobiology. J Neurosci. 2021 Sep 15;41(37):7698-7711. doi: 10.1523/JNEUROSCI.0619-21.2021. PMID 34526407